CLINICAL TRIAL: NCT00313352
Title: Effects of Beta-adrenergic Blocking Agents in Adult Patients With Transposition of the Great Arteries on Systemic Ventricular Function
Brief Title: Effects of Beta-adrenergic in Adults w/Transposition of Great Arteries on Systemic Ventricular Function
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Wendy M. Book, Principal Investigator, Emory University
Other Study IDs: 0293-2006
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Congenital Disorders
Keywords: adult; cardiac; transposition of great arteries; beta-adrenergic blockers
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Transposition of Great Vessels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this chart review study is to examine the effects of beta -adrenergic blocking agents on systemic ventricular dimensions, systemic atrioventricular valve function and exercise tolerance in patients with transposition of the great arteries (TGA) and systemic ventricular dysfunction.

DETAILED DESCRIPTION:
Many children with transposition of the great arteries who underwent atrial inflow correction using the Mustard or Senning operation are now adults. While their short- and midterm prognosis have been good, their life expectancy is limited by the onset of serious cardiovascular complications including arrhythmias, systemic (morphologically right) ventricular dysfunction and sudden cardiac death.

The ability of the morphological right ventricle (RV) to support the systemic circulation is limited. It has been postulated that perfusion and wall motion abnormalities are common in the systemic RV late (10-20 years) after Mustard's operation. Poor ventricular function causes progressive RV enlargement and systemic atrioventricular valve insufficiency, resulting in congestive heart failure (CHF). Deterioration in systolic function of the systemic ventricle is a major determinant of survival in these patients.

Little is known about the most effective therapy of progressive systemic RV dysfunction in these patients. Despite several recent studies demonstrating the benefit of beta-adrenergic blocking agents in improved left ventricular function in adults with heart failure and left ventricular dysfunction, there have been no reports of the use of beta-adrenergic blocking agents in adult patients with ventricular dysfunction due to congenital heart disease. This data collection study will be a single center, retrospective study; a chart review of patients with TGA (either DTGA or LTGA) and systemic right ventricular dysfunction.

Patient Population:

Patients followed-up at Emory University Hospital and The Emory Clinic who meet the following inclusion criteria:

1. Age ≥ 18 years
2. Diagnosis: Complete d-TGA or Congenitally Corrected TGA with a systemic morphologic right ventricle
3. Patients > 18 years of age seen at The Emory Clinic and Emory University Hospital with transposition of the great arteries
4. Systemic ventricular ejection fraction < 50% with or without a clinical diagnosis of heart failure
5. Echocardiogram performed between January 1, 1997and February 1, 2006

Future Directions:

The effects of beta-adrenergic blocking agents in patients with TGA and congestive heart failure due to systemic ventricular dysfunction have never been studied. To our knowledge, only one case report suggests that carvedilol may potentially improve systemic ventricular functions and volumes in these patients. This study will identify the potential merits of beta-blocker therapy in patients with TGA and CHF and could theoretically lead to a multi-institutional prospective analysis of beta-blocker therapy in adult patients with congenial heart disease and CHF.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed-up at Emory University Hospital and The Emory Clinic who meet the following inclusion criteria:

  1. Age ≥ 18 years
  2. Diagnosis: Complete d-TGA or Congenitally Corrected TGA with a systemic morphologic right ventricle
  3. Patients > 18 years of age seen at The Emory Clinic and Emory University Hospital with transposition of the great arteries
  4. Systemic ventricular ejection fraction < 50% with or without a clinical diagnosis of heart failure
  5. Echocardiogram performed between January 1, 1997and February 1, 2006

Exclusion Criteria:

* Those who do not meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective study analysis of medical records of patients age 18yrs and up, who had systemic RV dysfunction late after atrial inflow correction for d-TGA.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 1997-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
functional class | 6 months to 5 years
  beta blockers improved functional class in patient's with transposition and systemic right ventricles

CONTACTS AND LOCATIONS:
Overall Officials: Wendy M Book, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States